CLINICAL TRIAL: NCT00649389
Title: A Randomized, Double-Blind, Parallel Group Study Evaluating the Efficacy and Safety of Co-Administration of a Triple Combination Therapy of Olmesartan Medoxomil, Amlodipine Besylate and Hydrochlorothiazide in Subjects With Hypertension
Brief Title: Safety and Efficacy Study of a Triple Combination Therapy in Subjects With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Executive Director Clinical Development, Daiichi Sankyo Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS8635-A-U301
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2010-09-01 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2010-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- OM40/AML10 (Experimental): olmesartan medoxomil 40mg and amlodipine 10mg
  Interventions: Drug: Olmesartan medoxomil; Drug: Amlodipine
- OM40/HCTZ25 (Active Comparator): olmesartan medoxomil 40mg and hydrochlorothiazide 25mg
  Interventions: Drug: Olmesartan medoxomil; Drug: Hydrochlorothiazide
- AML10/HCTZ25 (Active Comparator): amlodipine 10mg and hydrochlorothiazide 25mg
  Interventions: Drug: Amlodipine; Drug: Hydrochlorothiazide
- OM40/AML10/HCTZ25 (Active Comparator): olmesartan medoxomil 40mg, amlodipine 10mg, and hydrochlorothiazide 25mg
  Interventions: Drug: Olmesartan medoxomil; Drug: Amlodipine; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Olmesartan medoxomil — 40mg olmesartan medoxomil
  Other Names: Benicar
  Arms: OM40/AML10; OM40/AML10/HCTZ25; OM40/HCTZ25
Drug: Amlodipine — Amlodipine 10mg
  Other Names: Norvasc
  Arms: AML10/HCTZ25; OM40/AML10; OM40/AML10/HCTZ25
Drug: Hydrochlorothiazide — Hydrochlorothiazide 25mg
  Arms: AML10/HCTZ25; OM40/AML10/HCTZ25; OM40/HCTZ25

SUMMARY:
To determine the effectiveness of four different strength combinations of three approved anti-hypertension therapies (olmesartan medoxomil, amlodipine, and hydrochlorothiazide) for lowering blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrable hypertension defined as mean sitting trough cuff blood pressure ≥ 140/100 mmHg (SeSBP ≥ 140 mmHg and SeDBP ≥ 100mmHg) or mean sitting trough cuff BP ≥ 160/90 mmHg (SeSBP ≥ 160 mmHg and SeDBP ≥ 90mmHg).
* Male or female newly diagnosed hypertensive subjects or currently on hypertension medication.

  * Negative urine pregnancy test at screening
  * Not lactating
  * Do not plan to become pregnant during the study
  * Will practice birth control throughout the study by the following: oral or patch contraceptive, injectable or implantable contraceptive medication, intrauterine device, diaphragm or female condom plus spermicide

    * Non childbearing potential must be classified by one of the following criteria
    * Had a hysterectomy or tubal ligation at least 6 months prior to consent
    * Has been postmenopausal for a least 1 year

Exclusion Criteria:

* Mean sitting trough cuff DBP <90 mmHg or mean sitting trough cuff SBP <140 mmHg (off antihypertensive medication).
* Subjects with uncontrolled hypertension taking multiple antihypertensive therapies (at the discretion of the investigator).
* Signs or symptoms which could exacerbate the occurrence of hypotension such as volume and salt depletion.
* History of hypertensive encephalopathy, stroke or transient ischemic attack (TIA).
* Participation in another clinical trial involving an investigational drug within one month prior to screening.
* History of myocardial infarction, percutaneous transluminal coronary revascularization, coronary artery bypass graft, and/or unstable angina within the past 6 months.
* Any history of New York Heart Association Class III or IV congestive heart failure (CHF). A history of New York Heart Association Class I or II CHF may be exclusionary at the discretion of the investigator.
* History of secondary hypertension including renal disease, pheochromocytoma, or Cushing's syndrome.
* Uncorrected coarctation of the aorta, bilateral renal artery stenosis, or unilateral renal artery stenosis in a solitary kidney.
* Evidence of symptomatic resting bradycardia.
* Evidence of hemodynamically significant cardiac valvular disease.
* Presence of heart block greater than first degree atrioventricular block, chronic atrial fibrillation or flutter.
* Uncontrolled Type I or Type II diabetes defined as HbA1c >9.0%. Diabetics must have documentation of HbA1c within 6 months of the Screening Visit. Undocumented subjects must have their HbA1c assessed prior to randomization. Note: Subjects with Type I or Type II diabetes controlled with insulin, diet or oral hypoglycemic agents on a stable dose for at least 30 days may be included.
* Evidence of liver disease as indicated by ALT and AST and/or total bilirubin >3 times the upper limit of normal.
* Severe renal insufficiency defined as a creatinine clearance (based on the Cockcroft-Gault formula) of <30 mL/min.
* Clinically significant laboratory elevations at Visit 1 that compromise subject safety, based on the investigator's judgment. Consideration should take into account the potential laboratory effects of the component blinded therapies.
* Positive for any one of the following tests: hepatitis B surface antigen, hepatitis C antibody (confirmed by radio immunobinding assay, RIBA) or HIV antibody (confirmed by western blot assay).
* Subjects with malignancy during the past 2 years excluding squamous cell or basal cell carcinoma of the skin.
* Known allergy to any of the medications used in the study.
* Subjects who require or are taking any concomitant medication, which may interfere with the objectives of the study (Refer to Section 5.2 for a listing of excluded medications).
* Pregnant or lactating females.
* Current history of drug or alcohol abuse.
* A subject with any medical condition, which in the judgment of the Investigator would jeopardize the evaluation of efficacy or safety and/or constitute a significant safety risk to the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (232):
- United States (228):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Gulf Shores, Alabama
  - Hoover, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Muscle Shoals, Alabama
  - Tuscumbia, Alabama
  - Chandler, Arizona
  - Goodyear, Arizona
  - Lake Havasu City, Arizona
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Searcy, Arkansas
  - Anaheim, California
  - Beverly Hills, California
  - Buena Park, California
  - Burbank, California
  - Carmichael, California
  - Chino, California
  - Chula Vista, California
  - Escondido, California
  - Greenbrae, California
  - Hollywood, California
  - Huntington Park, California
  - Long Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - Merced, California
  - National City, California
  - Orange, California
  - Roseville, California
  - San Diego, California
  - San Jose, California
  - Santa Ana, California
  - Santa Monica, California
  - Temecula, California
  - West Palm Beach, California
  - Westlake Village, California
  - Denver, Colorado
  - Golden, Colorado
  - Pueblo, Colorado
  - Wheat Ridge, Colorado
  - Danbury, Connecticut
  - Milford, Connecticut
  - Stamford, Connecticut
  - Trumbull, Connecticut
  - Waterbury, Connecticut
  - Aventura, Florida
  - Boynton Beach, Florida
  - Bradenton, Florida
  - Brooksville, Florida
  - Cape Coral, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Crystal River, Florida
  - Daytona Beach, Florida
  - Deerfield Beach, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - Dunnellon, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Largo, Florida
  - Merritt Island, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - West Bradenton, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Suwanee, Georgia
  - Waycross, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Libertyville, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Newton, Kansas
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Madisonville, Kentucky
  - Mount Sterling, Kentucky
  - Munfordville, Kentucky
  - Paducah, Kentucky
  - Kenner, Louisiana
  - Lake Charles, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Elkridge, Maryland
  - Oxon Hill, Maryland
  - Brockton, Massachusetts
  - Haverhill, Massachusetts
  - West Yarmouth, Massachusetts
  - Benzonia, Michigan
  - Clarkston, Michigan
  - Paw Paw, Michigan
  - Southfield, Michigan
  - Traverse City, Michigan
  - Waterford, Michigan
  - Brooklyn Center, Minnesota
  - Chaska, Minnesota
  - Saint Paul, Minnesota
  - Olive Branch, Mississippi
  - Florissant, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Butte, Montana
  - Missoula, Montana
  - Broken Bow, Nebraska
  - North Platte, Nebraska
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Elizabeth, New Jersey
  - Voorhees Township, New Jersey
  - Buffalo, New York
  - Manlius, New York
  - Mineola, New York
  - New York, New York
  - Westfield, New York
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Hickory, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Tabor City, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Austintown, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Euclid, Ohio
  - Franklin, Ohio
  - Kettering, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Mount Gilead, Ohio
  - Wadsworth, Ohio
  - Westlake, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Bensalem, Pennsylvania
  - Downingtown, Pennsylvania
  - Erie, Pennsylvania
  - Harleysville, Pennsylvania
  - Jenkintown, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Penndel, Pennsylvania
  - Philadelphia, Pennsylvania
  - Cranston, Rhode Island
  - East Providence, Rhode Island
  - Providence, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Murrells Inlet, South Carolina
  - Orangeburg, South Carolina
  - Rapid City, South Dakota
  - Bristol, Tennessee
  - Fayetteville, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - New Tazewell, Tennessee
  - Tullahoma, Tennessee
  - Austin, Texas
  - Bedford, Texas
  - Corpus Christi, Texas
  - Houston, Texas
  - Hurst, Texas
  - Lake Jackson, Texas
  - Midland, Texas
  - Plano, Texas
  - Round Rock, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Sugar Land, Texas
  - Temple, Texas
  - Waco, Texas
  - Bountiful, Utah
  - Magna, Utah
  - Midvale, Utah
  - Salt Lake City, Utah
  - Sandy City, Utah
  - Saratoga Springs, Utah
  - West Jordan, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Suffolk, Virginia
  - Federal Way, Washington
  - Lakewood, Washington
  - Tacoma, Washington
  - Kenosha, Wisconsin
  - Madison, Wisconsin
- Puerto Rico (4):
  - Ciales
  - Guayama
  - Ponce
  - Rio Piedras

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Kereiakes DJ, Chrysant SG, Izzo JL Jr, Littlejohn T 3rd, Melino M, Lee J, Fernandez V, Heyrman R. Olmesartan/amlodipine/hydrochlorothiazide in participants with hypertension and diabetes, chronic kidney disease, or chronic cardiovascular disease: a subanalysis of the multicenter, randomized, double-blind, parallel-group TRINITY study. Cardiovasc Diabetol. 2012 Oct 30;11:134. doi: 10.1186/1475-2840-11-134. PMID 23110471
- [Derived] Chrysant SG, Littlejohn T 3rd, Izzo JL Jr, Kereiakes DJ, Oparil S, Melino M, Lee J, Fernandez V, Heyrman R. Triple-Combination therapy with olmesartan, amlodipine, and hydrochlorothiazide in black and non-black study participants with hypertension: the TRINITY randomized, double-blind, 12-week, parallel-group study. Am J Cardiovasc Drugs. 2012 Aug 1;12(4):233-43. doi: 10.1007/BF03261832. PMID 22799613
- [Derived] Oparil S, Melino M, Lee J, Fernandez V, Heyrman R. Triple therapy with olmesartan medoxomil, amlodipine besylate, and hydrochlorothiazide in adult patients with hypertension: The TRINITY multicenter, randomized, double-blind, 12-week, parallel-group study. Clin Ther. 2010 Jul;32(7):1252-69. doi: 10.1016/j.clinthera.2010.07.008. PMID 20678674
- [Derived] Chrysant SG, Oparil S, Melino M, Karki S, Lee J, Heyrman R. Efficacy and safety of long-term treatment with the combination of amlodipine besylate and olmesartan medoxomil in patients with hypertension. J Clin Hypertens (Greenwich). 2009 Sep;11(9):475-82. doi: 10.1111/j.1751-7176.2009.00159.x. PMID 19751459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit 12 May 2008. Last subject last follow-up 27 Feb 2009. 317 sites in USA and Puerto Rico. Planned: 2400 subjects (600 per treatment arm). Enrolled: 6724 subjects. Randomized: 2492 subjects.
Pre-assignment Details: Duration of the study was 57 weeks with 52 weeks of treatment. This included 3-week stabilization/washout (Period I), 12-week double blind treatment (Period II), 40 week open label treatment (Period III), and 2-week post treatment follow-up (Period IV).
Groups:
- OM40/AML10: Double blind treatment olmesartan medoxomil (OM) 40 mg, Amlodipine (AML) 10 mg tablets once daily.
- OM40/HCTZ25: Double blind treatment olmesartan medoxomil (OM) 40 mg, Hydrochlorothiazide (HCTZ) 25 mg tablets once daily.
- AML10/HCTZ25: Double blind treatment Amlodipine (AML) 10 mg, Hydrochlorothiazide (HCTZ) 25 mg tablets once daily.
- OM40/AML10/HCTZ25: Double blind treatment olmesartan medoxomil (OM) 40 mg, Amlodipine (AML) 10 mg, Hydrochlorothiazide (HCTZ) 25 mg, tablets once daily.
Period: Overall Study
Arm/Group | OM40/AML10 | OM40/HCTZ25 | AML10/HCTZ25 | OM40/AML10/HCTZ25
Started | 628 | 637 | 600 | 627
Completed | 557 | 531 | 512 | 516
Not Completed | 71 | 106 | 88 | 111
Not completed — Adverse Event | 22 | 46 | 38 | 48
Not completed — Lost to Follow-up | 15 | 17 | 21 | 26
Not completed — Protocol Violation | 11 | 13 | 9 | 8
Not completed — Withdrawal by Subject | 20 | 21 | 19 | 23
Not completed — Other | 3 | 9 | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OM40/AML10 | OM40/HCTZ25 | AML10/HCTZ25 | OM40/AML10/HCTZ25 | Total
Number analyzed (Participants) | 628 | 637 | 600 | 627 | 2492
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 508 | 505 | 504 | 504 | 2021
  >=65 years | 120 | 132 | 96 | 123 | 471
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.93) | 55.9 (10.78) | 54.6 (10.82) | 54.7 (11.22) | 55.1 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303 | 298 | 266 | 307 | 1174
  Male | 325 | 339 | 334 | 320 | 1318
Race/Ethnicity, Customized [Number; unit: Participants] — Race of participants as selected by participant. Participants were allowed to choose more than one race category; therefore, the total for an arm may be greater than the number of participants
  Participants
    American Indian/Alaskan Native | 3 | 1 | 4 | 1 | 9
    Asian | 13 | 10 | 7 | 19 | 49
    Hawaiian/Pacific Islander | 0 | 1 | 1 | 2 | 4
    Black/African American | 181 | 200 | 192 | 184 | 757
    White | 431 | 421 | 391 | 415 | 1658
    Unknown or Not Reported | 0 | 4 | 5 | 6 | 15
Diabetes Status [Number; unit: Participants]
  Diabetic | 100 | 99 | 92 | 96 | 387
  Not diabetic | 528 | 538 | 508 | 531 | 2105
Weight [Mean (Standard Deviation); unit: kg] | 95.9 (22.65) | 96.1 (22.55) | 96.1 (23.41) | 96.0 (23.24) | 96.0 (22.94)
Body Mass Index [Number; unit: Participants]
  Less than 30 kg/m2 | 229 | 238 | 230 | 240 | 937
  Greater than or equal to 30 kg/m2 | 399 | 399 | 370 | 387 | 1555
Duration of hypertension [Mean (Standard Deviation); unit: years] | 10.12 (9.865) | 10.34 (9.826) | 9.73 (8.983) | 9.54 (9.558) | 9.94 (9.571)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Seated Diastolic Blood Pressure (SeDBP).
Time Frame: baseline to 12 weeks
Population: The full analysis set consists of subjects who received at least 1 dose of study medication and had a baseline and at least one post-dose assessment of SeDBP
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM40/AML10 | OM40/HCTZ25 | AML10/HCTZ25 | OM40/AML10/HCTZ25
Number analyzed (Participants) | 624 | 627 | 593 | 614
mm Hg | -17.8 (9.47) | -16.5 (10.84) | -14.8 (8.78) | -21.5 (10.25)
Statistical Analysis 1: Comparison: OM40/AML10 vs OM40/AML10/HCTZ25; All treatment comparisons were calculated as OM40/AML10/HCTZ25 minus the respective dual combination treatment group. Least-squares mean differences, SEs, and 2-sided p-values were obtained from an ANCOVA model with baseline blood pressure as a covariate, and fixed effects of treatment, age group, race group, and diabetic status; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: OM40/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: AML10/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Percentage of Subjects Who Reached Blood Pressure Goal (<140/90 mmHg; <130/80 mmHg for Subjects With Diabetes, Chronic Renal Disease, or Chronic Cardiovascular Disease)by 12 Weeks
Time Frame: Baseline to 12 weeks
Population: The full analysis set consists of subjects who received at least 1 dose of study medication and had a baseline and at least one post-dose assessment of seated diastolic blood pressure
Measure: Number; unit: Percentage of subjects
Arm/Group | OM40/AML10 | OM40/HCTZ25 | AML10/HCTZ25 | OM40/AML10/HCTZ25
Number analyzed (Participants) | 624 | 627 | 593 | 614
Percentage of subjects | 46.0 | 46.6 | 34.9 | 64.3
Statistical Analysis 1: Comparison: OM40/AML10 vs OM40/AML10/HCTZ25; Each p-value was obtained from individual Cochran-Mantel-Haenszel tests stratified by age group, race group, and diabetic status comparing the triple combination therapy to each dual combination; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: OM40/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: AML10/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change in Mean 24-hour Ambulatory Blood Pressure From Baseline to Week 12 or Early Termination
Time Frame: Baseline to 12 weeks or early termination
Population: The ABPM Analysis Set included 440 subjects who provided consent to participate in the ABPM sub-study and who were to provide ABPM measurements prior to and after randomization. Those analyzed is the number who had values at both baseline and 12 weeks or early termination
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM40/AML10 | OM40/HCTZ25 | AML10/HCTZ25 | OM40/AML10/HCTZ25
Number analyzed (Participants) | 96 | 101 | 83 | 100
mm Hg
  Diastolic blood pressure | -13.9 (8.09) | -14.5 (8.73) | -10.7 (7.46) | -18.0 (8.11)
  Systolic blood pressure | -23.5 (11.80) | -23.9 (13.10) | -18.5 (10.67) | -30.3 (13.85)
Statistical Analysis 1: Comparison: OM40/AML10 vs OM40/AML10/HCTZ25; Diastolic blood pressure: All treatment comparisons were calculated as OM40/AML10/HCTZ25 minus the respective dual combination treatment group. Least-squares mean differences, SEs, and 2-sided p-values were obtained from an ANCOVA model with baseline blood pressure as a covariate, and fixed effects of treatment, age group, race group, and diabetic status; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: OM40/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: AML10/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA
Statistical Analysis 4: Comparison: OM40/AML10 vs OM40/AML10/HCTZ25; Systolic blood pressure: All treatment comparisons were calculated as OM40/AML10/HCTZ25 minus the respective dual combination treatment group. Least-squares mean differences, SEs, and 2-sided p-values were obtained from an ANCOVA model with baseline blood pressure as a covariate, and fixed effects of treatment, age group, race group, and diabetic status; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: OM40/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 6: Comparison: AML10/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p < 0.0001, ANCOVA

4. Secondary Outcome: Change in Seated Systolic Blood Pressure From Baseline to Week 12
Time Frame: Baseline to week 12
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM40/AML10 | OM40/HCTZ25 | AML10/HCTZ25 | OM40/AML10/HCTZ25
Number analyzed (Participants) | 624 | 627 | 593 | 614
mm Hg | -31.1 (15.44) | -31.2 (18.58) | -28.9 (15.12) | -38.1 (17.40)
Statistical Analysis 1: Comparison: OM40/AML10 vs OM40/AML10/HCTZ25; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: OM40/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: AML10/HCTZ25 vs OM40/AML10/HCTZ25; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety was assessed at all study visits. Variables included adverse events, clinical laboratory tests, vital signs, ECGs, and physical examinations. The assessment of causality was based on the investigator's judgment.
Arm/Group | OM40/AML10 | OM40/HCTZ25 | AML10/HCTZ25 | OM40/AML10/HCTZ25
Serious Adverse Events (participants affected / at risk) | 9/596 | 7/580 | 9/552 | 10/574
Other Adverse Events (participants affected / at risk) | 210/596 | 210/580 | 212/552 | 237/574
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OM40/AML10 (N=596) | OM40/HCTZ25 (N=580) | AML10/HCTZ25 (N=552) | OM40/AML10/HCTZ25 (N=574)
appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
sepsis (Infections and infestations) | 0 | 0 | 1 | 0
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
cerebrovasular accident (Nervous system disorders) | 0 | 2 | 0 | 0
ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
cerebellar infarction (Nervous system disorders) | 0 | 1 | 0 | 0
hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1
syncope (Nervous system disorders) | 0 | 0 | 0 | 1
coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 2
acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
gastrointstial haemhorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
rectal haemhorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1
fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
vertebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
pulmonary artery atresia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OM40/AML10 (N=596) | OM40/HCTZ25 (N=580) | AML10/HCTZ25 (N=552) | OM40/AML10/HCTZ25 (N=574)
dizziness (Nervous system disorders) | 29 | 58 | 17 | 57
headache (Nervous system disorders) | 42 | 38 | 33 | 37
upper respiratory tract infection (Infections and infestations) | 26 | 18 | 14 | 16
nasopharyngitis (Infections and infestations) | 11 | 20 | 16 | 20
edema peripheral (General disorders) | 42 | 6 | 46 | 44
fatigue (General disorders) | 34 | 31 | 36 | 24
muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 14 | 13 | 18
nausea (Gastrointestinal disorders) | 12 | 22 | 12 | 17
hypokalemia (Metabolism and nutrition disorders) | 2 | 3 | 25 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study site may not publish results of study until after coordinated multicenter publication has been submitted for publication or one year after study has ended, whichever occurs first. Therefore, study site will have the opportunity to publish results of study, provided that Daiichi Sankyo has had the opportunity to review and comment on study site's proposed publication prior to being submitted for publication with advice of company patent council and in accord with subject protection needs.